CLINICAL TRIAL: NCT07267533
Title: Precise 3D Surview Clinical Study
Brief Title: Precise 3D Surview
Acronym: 3D Surview
Status: Not yet recruiting | Type: Observational
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Collaborators: Philips Healthcare (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: Precise 3D Surview
Record Dates: First submitted 2025-09-23; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-09

CONDITIONS: Computed Tomography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

SUMMARY:
The purpose of the study is to assess the performance of Precise 3D Surview on CT 5300 and Incisive CT Scanners as compared with manual annotation by experienced CT technologists.

* To evaluate the acceptance rate of the Auto 3D Planning Box compared with manual annotation by experienced CT technologists.
* To evaluate the acceptance rate of the Auto Suggestion for Locator compared with manual annotation by experienced CT technologists.
* To evaluate the acceptance rate of the Auto Planning for Truncated Anatomies (lung and liver) compared with manual annotation by experienced CT technologists.
* To evaluate the acceptance rate of Auto Planning and Symmetry Correction for Tilted Head compared with manual annotation by experienced CT technologists.

ELIGIBILITY:
Inclusion Criteria:

* Subjects scanned by CT 5300 (K232491) and Incisive CT (K212441) according to the department standard of care clinical protocols.
* Subjects age is over eighteen (18) years1.
* Patients scanned in supine orientation.
* Non-contrast CT scan
* CT scan with standard resolution

Exclusion Criteria:

* Subjects age is under or equal 18 years old
* Patients are not scanned in supine orientation.
* Contrast-enhanced CT scans.
* CT scans with high resolution
* Scans that are not completed due to technical difficulties

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults
Sampling Method: Probability Sample
Enrollment: 274 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Acceptance rate of the 3D Surview | Reading session at 4 months